CLINICAL TRIAL: NCT06955026
Title: Effect of the Hockey Slideboard Training Combined With Blood Flow Restriction (BFR) in the Rehabilitation Following Anterior Cruciate Ligament Surgical Reconstruction (ACL-R)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spitalul Municipal Odorheiu Secuiesc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOCT1
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Anterior Cruciate Ligament Rupture; Rehabilitation After ACL Reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL-R with hockey slideboard training combined with blood flow restriction (BFR) (Experimental): Patients underwent ACL-R who undergo a reathletization program as usual together with the use of the hockey slideboard combined with BFR training
  Interventions: Other: Hockey slideboard combined with BFR training
- ACL-R with hockey slideboard training (Active Comparator): Patients underwent ACL-R who undergo a reathletization program as usual together with the use of the hockey slideboard
  Interventions: Other: Hockey slideboard

INTERVENTIONS:
Other: Hockey slideboard combined with BFR training — Hockey slideboard combined with BFR training
  Arms: ACL-R with hockey slideboard training combined with blood flow restriction (BFR)
Other: Hockey slideboard — Hockey slideboard
  Arms: ACL-R with hockey slideboard training

SUMMARY:
ACL injuries represent a major health and economic burden. The overall incidence of ACL injuries has increased and is likely to continue to increase, in part due to increased sports participation.

In the acute post-surgical phase there is a period of physiologic recovery from the surgical injury and subsequent relative muscle disuse that is associated with atrophy loss of strength and anterior knee pain. Therefore, improvement of muscle function is a priority in the rehabilitation and reathletization process.

To achieve significant muscle hypertrophy as well as a possible subsequent increase in strength, it is widely accepted that resistance exercises with relevant load (~70% of the one repetition maximum - 1RM) are necessary; however, in patients undergoing anterior cruciate ligament reconstruction (ACL-R), exercises with high loads are considered unsafe in the early stages and could increase the risk of re-injury.

BFR training is an established muscle training and rehabilitation technique in which the blood supply to and from the muscles involved in the exercise is restricted using an external device.

Although the physiological mechanisms related to this intervention are not yet well understood, it is thought that in BFR training, despite the low level of mechanical tension, the main driver of myocellular hypertrophy could be metabolic stress that is realized by local accumulation of metabolites. Thus, it seems that hypertrophic adaptations can be induced with much lower exercise intensities using BFR. In fact, when combined with low-load resistance training (e.g., 20% 1RM), training with BFR has shown positive results in increasing muscle volume and strength after ACL-R in complete safety comparable to standard training without BFR.

It has also already been demonstrated how incorporating the use of the hockey slideboard into the rehabilitation procedure following ACL-R gives benefits in terms of strength recovery of the extensor muscles of the operated limb with the same safety profiles as standard rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* having undergone ACL-R following a unilateral rupture, with reconstructive surgical technique by bone-patellar tendon-bone autograft (BPTB) or semitendinosus-gracilis autograft (STG)
* ACL-R including associated meniscal lesions treated with selective meniscectomy and/or non-complex meniscal suture

Exclusion Criteria:

* not having undergone ACL-R following a unilateral rupture, with reconstructive surgical technique by bone-patellar tendon-bone autograft (BPTB) or semitendinosus-gracilis autograft (STG)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Adductor muscles maximal voluntary isometric contraction (MVIC) | Before the study intervention (T0) and after the study intervention lasting for four weeks (T1)
  Adductor muscles' maximal voluntary isometric contraction (MVIC) measured via hand-held dynamometer test in a supine position

SECONDARY OUTCOMES:
Abductor muscles maximal voluntary isometric contraction (MVIC) | Before the study intervention (T0) and after the study intervention lasting for four weeks (T1)
  Abductor muscles' maximal voluntary isometric contraction (MVIC) measured via hand-held dynamometer test in a supine position
Adductor/abductor isometric strength (MVIC) ratio | Before the study intervention (T0) and after the study intervention lasting for four weeks (T1)
  Adductor and abductor muscles' maximal voluntary isometric (MVIC) strength ratio measured via hand-held dynamometer test in a supine position
Y-balance test (YBT) composite score | Before the study intervention (T0) and after the study intervention lasting for four weeks (T1)
  The YBT assessment demands that the athlete maintain balance on one leg while extending the opposite leg as far as feasible in three different directions: anterior, posterolateral, and posteromedial. The YBT composite score is calculated by summing the three reach distances and normalizing them to the lower limb length.
Triple hop test for distance | After the study intervention lasting for four weeks (T1)
  Triple hop test executed, calculating the maximum reached distance and comparing the healthy limb result with the involved leg.
Single hop test for distance | After the study intervention lasting for four weeks (T1)
  Single hop test executed, calculating the maximum reached distance and comparing the healthy limb result with the involved leg.
Side hop test | After the study intervention lasting for four weeks (T1)
  The participant is required to hop from side to side on one limb outside two parallel strips of tape 40 cm apart, and instructed to hop as many hops as possible for 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Spital Municipal Odorheiu Secuiesc, Odorheiu Secuiesc, Romania, Romania

IPD SHARING:
Plan to Share IPD: No